CLINICAL TRIAL: NCT05979272
Title: Development and Preliminary Testing of an Adjunct Smartphone App to Reduce Marijuana Use in Court-Involved, Non-Incarcerated Adolescents
Brief Title: TECH App Marijuana Use Intervention for Court-Involved Adolescents
Acronym: TECH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Brown University (Other); Rhode Island Hospital (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Sarah Helseth, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SP0078326; K23DA048062 (NIH)
Record Dates: First submitted 2023-07-31; First posted 2023-08-07 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Cannabis Use; Adolescent
Keywords: Court-involved; cannabis use; adolescent; marijuana use; digital health; mHealth; smartphone; juvenile justice; juvenile legal
MeSH Terms: conditions — Marijuana Use | interventions — Therapeutics; PLEKHG5 protein, human; Amyloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TAU-only (Active Comparator): Treatment as usual
  Interventions: Behavioral: Treatment as usual
- TAU + TECH (Experimental): Treatment as usual, plus TECH app
  Interventions: Behavioral: Treatment as usual; Behavioral: Teen Empowerment through Computerized Health (TECH) app

INTERVENTIONS:
Behavioral: Treatment as usual — Treatment as Usual at the local family court, which includes a brief, computerized motivation enhancement intervention. All CINI youth will receive TAU, regardless of condition.
Behavioral: Teen Empowerment through Computerized Health (TECH) app — An adjunct smartphone app (i.e., TECH) developed to support TAU. All participants randomly assigned to TAU+TECH will receive the TECH app.
  Arms: TAU + TECH

SUMMARY:
The study is about helping teens who are involved in the court system to cut down or quit using marijuana. Teens may be asked to test out an experimental smartphone app, called TECH, that will be used only by teens in this study. This app is a private online community where teens can work towards changing their substance use and other behavior with the help of other anonymous teens. We will use this information to learn how the app may help teens make a change and to improve the TECH app.

DETAILED DESCRIPTION:
This multiphase study will establish the feasibility, acceptability, and preliminary efficacy of a novel smartphone app that leverages both intrapersonal and interpersonal mechanisms to promote cannabis-related behavior change among CINI youth ages 14-17. The app, Teen Empowerment through Computerized Health (TECH), will be evaluated as an adjunct to treatment as usual (TAU) at the local family court. Phase 1 (completed Fall 2021) included a series of semi-structured interviews with key individuals, to inform how clinical goals (e.g., reduced cannabis use) will map onto usage goals (e.g., goal-setting, peer networking), features (e.g., expert-moderated forum, notifications) and workflow. Then, Phase 2 (completed Fall 2022) beta tested and iteratively refined the TECH prototype with 10 court-involved, non-incarcerated (CINI) youth. In the current phase of the work, Phase 3, we will conduct a pilot randomized control trial (RCT) with 60 CINI youth to test the TECH app (TAU+TECH) relative to TAU-only.

Specific aims are:

Aim 1. Apply the Behavior Intervention Theory model to develop a user-driven tool (i.e., TECH) that capitalizes on how, why, and when CINI youth would most prefer to engage with a smartphone app to reduce cannabis use.

~Aim 1 was achieved in Phase 1 qualitative interviews with CINI youth, their parents, and behavioral health app developers.

Aim 2. Examine the feasibility and acceptability of the TECH user-driven smartphone app.

~Hypothesis 1 is that TECH will be feasible and acceptable to CINI youth, as measured via enrollment and withdrawal rates, app usage data, and exit interviews. Aim 2 will be achieved through Phase 2 beta testing (n = 10) and Phase 3's pilot RCT (n = 60) with CINI youth.

Aim 3. Test the preliminary efficacy of the TECH smartphone app as an adjunct to TAU (TECH + TAU vs. TAU-only) on cannabis use (primary outcome).

~Hypothesis 2 is that, relative to CINI youth who receive TAU-only, the TAU+TECH group will demonstrate greater reductions in cannabis use. Aim 3 will be achieved via Phase 3's pilot RCT (n = 60 CINI youth).

ELIGIBILITY:
Inclusion Criteria:

* Aged 14 years to 18 years
* Able to speak and read English
* Have access to a smartphone
* Self-report past-year cannabis use
* If a minor, able to provide parental consent and child assent

Exclusion Criteria for all participants is limited to conditions that would preclude active participation in an intervention study of a mobile app (e.g., psychosis, cognitive impairment, visual impairment).

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in days of cannabis use (Preliminary Efficacy) | Last 90 days at baseline, and 1-, 3-, and 6-months
  Self-report of total days of cannabis use, via Timeline Followback Interview

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Rhode Island Hospital, Chicago, Illinois
  - Rhode Island Family Court, Providence, Rhode Island
  - Brown University, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Helseth SA, Guigayoma J, Price D, Spirito A, Clark MA, Barnett NP, Becker SJ. Developing a Smartphone-Based Adjunct Intervention to Reduce Cannabis Use Among Juvenile Justice-Involved Adolescents: Protocol for a Multiphase Study. JMIR Res Protoc. 2022 Mar 11;11(3):e35402. doi: 10.2196/35402. PMID 35275086